CLINICAL TRIAL: NCT06953804
Title: Optimal Implementation of Antimicrobial Stewardship in General Practice (OPTIMAS-GP) Study: A Hybrid Type 3 Implementation Trial
Brief Title: Optimal Implementation of Antimicrobial Stewardship in General Practice
Acronym: OPTIMAS-GP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wollongong (Other)
Responsible Party: Principal Investigator, Andrew Bonney, Professor of General Practice, University of Wollongong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2024/337; MRFF project 2029531 (Other Grant/Funding Number: NHMRC); U1111-1319-2201 (Other: WHO)
Record Dates: First submitted 2025-04-07; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: The Use of Antimicrobial Stewardship in in General Practice (Family Medicine); Respiratory Tract Infections (RTI)
Keywords: hybrid type 3 implementation trial; cluster randomised control trial; antimicrobial stewardship; antibiotic stewardship; respiratory tract infections; general practice; family medicine; primary care; Australia
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Virtual network activities (Experimental): Participants randomised to the Virtual arm will receive online self-paced education modules regarding antimicrobial interventions, guided self-audit and reflection regarding intervention use, and reinforcement podcasts (~7 hours).
  Interventions: Other: Antimicrobial stewardship activities delivered through Virtual Network
- Integrated network activities (Experimental): Participants randomised to the Integrated Network arm will receive antimicrobial intervention education delivered by live interactive online webinar-based sessions, peer-group audit and reflection, and reinforcement online forum participation.
  Interventions: Other: Antimicrobial stewardship activities delivered through Integrated Network activities

INTERVENTIONS:
Other: Antimicrobial stewardship activities delivered through Virtual Network — Participants will receive online self-paced education modules regarding antimicrobial interventions, guided self-audit and reflection regarding intervention use, and reinforcement podcasts (~7 hours).
  Participants in the Virtual Newtwork arm will primarily receive these interventions online.
  Arms: Virtual network activities
Other: Antimicrobial stewardship activities delivered through Integrated Network activities — Participants will receive online self-paced education modules regarding antimicrobial interventions, guided self-audit and reflection regarding intervention use, and reinforcement podcasts (~7 hours).
  Participants in the Integrated Network arm will primarily receive these interventions face-to-face and active online activities.
  Arms: Integrated network activities

SUMMARY:
This trial aims to increase the use of antimicrobial stewardship resources when treating patients with respiratory tract infections. This trial is set in Australian general practices (family medicine or primary care).

The main question it aims to answer is which type of implementation activities increase the use of antimicrobial stewardship resources. Researchers will compare doctors who receive face-to-face implementation activities (the Integrated Network group) to those who received virtual or online activities (the Virtual Network group). The primary hypothesis is that there will be a difference in how often interventions are used

Participating doctors will be asked to record how often they use antimicrobial stewardship resources and which interventions they prefer. Participating practices will also provide researchers data on how many patients the doctors see.

Patients with respiratory tract infections who saw a participating doctor will be asked to give feedback on their experience using surveys. A subgroup of doctors, practice staff, and patients will interviewed about their experience in the study.

DETAILED DESCRIPTION:
SUMMARY The OptimasGP study is a two-arm superiority cluster-randomised Hybrid type 3 pragmatic implementation trial to promote the use of antimicrobial stewardship (AMS) interventions by doctors in general practice treating adults with respiratory tract infections.

The implementation strategies used in the trial will be delivered using a Virtual Network (arm 1) and Integrated Network (arm 2) approach. Data collection will collected for five months during winter for the baseline period, followed by implementation activities, and five months in the following winter post-activities.

The primary study outcome is AMS intervention use per 100 consultations. Secondary objectives are based on the RE-AIM framework for reach, efficacy, implementation, adoption, and maintenance of the implementation.

SETTING The study sites for the implementation study comprise 40 general practices across New South Wales, Queensland, Tasmania, and Victoria in Australia.

PARTICIPANTS Participants include 120 general practice (family practice) doctors, 40 practice staff, and patients with respiratory tract infections. Informed consent will be obtained from participating doctors and practice staff in written form by members of the research team. Approximately half of participants will be recruited in 2025, with the remainder recruited in 2026.

Patients will be sent invitations to participate in the study by practice staff via SMS. For patient surveys, completion of surveys will constitute tacit consent. For patients in the case-studies sub-group, informed consent will be obtained in written form by members of the research team.

There are two subgroups. In the first subgroup, three sites from each arm will be elected for the nested case-study (individual semi-structured interviews). For each site, interviewers will construct case studies consisting of 6-8 participants (e.g., 2 doctors, 1-2 practice nurses, 1 practice manager, and 4 ARI patients per case).

In the second subgroup, 3 sites per arm (6-9 doctors) will be provided with FebriDx point of care tests to identify if respiratory tract infections are bacterial or viral in origin. These tests have been approved by the USA FDA (K230917) and by the Australian Therapeutic Goods Administration (ref 346636).

Recruitment and retention will be facilitated by payments to participants.

INTERVENTION RESOURCES Participating doctors will be provided AMS interventions in an online AMS Toolbox (see the latest version at https://redcap.uow.edu.au/redcap/surveys/?s=37HKC3KFMLED7PY7) which they may use when treating eligible patients. The Toolbox will contain AMS interventions resource for shared decision-making between doctors and patients, delayed prescribing, and clinical decision support (including guidance for using FebriDx point of care devices for relevant members of the subgroup).

IMPLEMENTATION ACTIVITIES Both arms will complete ~7 hours of implementation activities. These activities will be provided by MedCast, an established provider of ongoing health professional education in Australia.

Participants in the Virtual arm will receive online self-paced education modules, guided self-audit and reflection regarding antimicrobial stewardship and use of AMS Toolbox components, and reinforcement podcasts.

Participants randomised to the Integrated Network arm will receive education delivered by live interactive online webinar-based sessions, peer-group audit and reflection, and reinforcement online forum participation.

DATA COLLECTION Doctors complete data entry using the AMS Toolbox by selecting if they used an intervention, which intervention was used, and whether an antibiotic was prescribed for immediate use, delayed use, or not prescribed. In addition, the number of patients seen by each doctor will be collected based on a fortnightly record of practice records using surveys.

Demographic data will be collected using online surveys.

Patients will completed patient-reported outcome measures and patient reported experience measures using online surveys. Interviews of the nested-case study sub-group will be qualitative in nature.

All surveys will using REDCap (Research Electronic Data Capture) forms hosted at the University of Wollongong.

RISKS As this study has a low risk of harm or death, and as no interim analyses are planned, the study will not have a Data Safety Monitoring Board. Harms will be recorded through PROMs and direct reports from participating doctors. Harms such as re-consultations and hospitalizations reported to the research team will be discussed with an independent data monitor. This monitor can cease the study at any time if concerns arise. No interim analysis is planned and thus no stopping guidelines are provided.

ELIGIBILITY:
Study sites

Inclusion Criteria:

1. New South Wales, Queensland, Tasmania, or Victoria
2. at least two GPs per practice consent to be in the study,
3. that at least one member of practice staff consents to be in the study
4. that a staff member from the site will be available to provide 90 minutes per fortnight of administrative support for the study. There are no exclusion criteria in addition to this.

Exclusion Criteria: None

Participating doctors and healthcare workers

Inclusion criteria:

1) Working at a participating practice for at least three days a week. Exclusion criteria : None

Patients completing patient reported outcome measure survey

Inclusion criteria:

1. patients consulted with a participating GP for a RTI,
2. patients re-consulted with a GP or was hospitalized. Exclusion criteria: None

Patient reported experience measures survey

Inclusion criteria:

1) patient consulted with a participating GP for an RTI. Exclusion criteria: None

Patients participating in interviews as part of the nested case studies

Inclusion criteria:

1. consulted with a participating GP for a RTI,
2. completed a patient survey,
3. able to read and speak English Exclusion criteria: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in use of antimicrobial interventions per 100 consults | From baseline for 5 months, from post intervention for 5 months
  This score is derived from the number of times an intervention is used (measured using the AMS Toolbox online form) divided by the number of participants a doctor sees (measured using an audit). Measuring periods are fortnightly.
  The eligible range is 0-100, with higher values indicating a better outcome.

SECONDARY OUTCOMES:
Reach: Number enrolled - Doctors | Enrolment
  Enrolment
  Enrolment rates of doctors will be determined for doctors by the number of online consents completed via Redcap. Higher numbers indicate better outcomes.
Reach: Representativeness of practices | Baseline
  A survey of practice size and location will be conducted.
Reach: Completions - Doctors | 5 months post intervention
  Completion rates of doctors will be determined by recording participant completion rates across all phases of the trial.
Reach: Representativeness of participating doctors and staff | Baseline.
  A survey of participating doctors and staff will be conducted to measure demographic and workplace variables.
Reach: Representativeness of patients | From baseline up to 5 months, from post intervention up 5 months
  Brief demographic questions will be asked of patients completing online surveys.
Effectiveness: Change in intervention use per 100 RTI consults | From baseline for 5 months, from post intervention for 5 months
  This score is derived from the number of times an intervention is used (measured using the AMS Toolbox online form) divided by the number of patients with a respiratory tract infection (RTI) a doctor sees (measured using an audit). Measuring periods are fortnightly. The eligible range is 0-100, with higher values indicating a better outcome.
Effectiveness: Change in antibiotics prescribed per 100 RTI consults | From baseline for 5 months, from post intervention for 5 months
  This score is derived from the number of times an antibiotic is prescribed (measured using the AMS Toolbox online form) divided by the number of patients with a respiratory tract infection (RTI) a doctor sees (measured using an audit). Measuring periods are fortnightly. The eligible range is 0-100, with higher values indicating a worse outcome.
Effectiveness: Change in antibiotic prescriptions given for RTIs (self-report) | From baseline for 5 months, from post intervention for 5 months
  This score is derived from the number of times an antibiotic is dispensed (measured using the AMS Toolbox online form) divided by the number of patients with an RTI a doctor sees (measured using AMS Toolbox). The eligible range is 0-100, with higher values indicating a worse outcome.
Effectiveness: Total antibiotics prescribed per 100 consults | From baseline for 5 months, from post intervention for 5 months
  This score is derived from the total number of times an antibiotic is prescribed (measured using the AMS Toolbox online form) per consults with patients.
  The eligible range is 0-100, with lower values indicating a better outcome.
Effectiveness: Adverse events | From baseline up to 5 months, from post intervention up 5 months
  An adverse event is defined as a reconsult with a participating doctor or hospitalisation related to an acute respiratory tract infection or related medical problems within 30 days of the initial consultation (measured through a patient-reported outcome measure), calculated by the total number of adverse events reported by patients.
Implementation: Fidelity to protocol during the study | 5 months post-intervention
  Fidelity will be measured qualitatively (using case study interviews) with participating doctors.
Implementation: Doctor experiences of interventions and implementation strategies | 5 months post baseline, 5 months post intervention
  User experiences will be measured qualitatively (using case study interviews), with participating doctors.
Implementation: Practice staffs' experiences of interventions and implementation strategies | 5 months post baseline, 5 months post intervention
  User experiences will be measured qualitatively (using case study interviews) with practice staff.
Implementation: Patients' experience of interventions and implementation strategies (qualitative) | 5 months post baseline, 5 months post intervention
  User experiences will be measured qualitatively (using case study interviews) with patients.
Implementation: Change in patients' experience of interventions and implementation strategies (quantitative) | From baseline up to 5 months, from post intervention up 5 months
  Patient-reported experience measure survey will be offered to eligible patients consulting with a participating GP. Surveys include seven questions each scored from 1-4 with higher outcomes worse. The eligible range is 7-28, with higher values indicating a worse outcome.
Adoption: Completion of implementation modules | Following the 5 months baseline period, and throughout the 5 months post intervention period.
  Completion of implementation activity modules will be tracked using data supplied by MedCast.
Adoption: Change in the use of individual AMS interventions | From baseline for 5 months, from post intervention for 5 months
  This score is derived from the number of times an intervention is used (measured using the AMS Toolbox online form) Toolbox) per 100 consults.
  The eligible range is 0-100, with higher values indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Bonney, PhD,, Principal Investigator — Graduate School of Medicine, University of Wollongong

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared in-deidentified form.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: For IPD, data will be available from December 2029.
  For supporting information, the protocol paper and statistical analysis plan will be submitted for publication by November 2025. Informed consent form is attached. Analytical code will be provided with the primary outcomes publication.
  IPD and supporting data will be available at least until December 2039.
Access Criteria: IPD:
  Supporting evidence: the protocol will be published in a peer-reviewed journal. Informed consent forms are available on request from the primary investigator or from the study website ().
  Analytical code will be provided with the primary outcomes publication

REFERENCES:
- See also: Study website — https://www.uow.edu.au/science-medicine-health/schools-entities/gsm/research/optimas-gp/
- See also: FDA approval of FebriDx for use in the USA — https://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfpmn/pmn.cfm?ID=K230917